CLINICAL TRIAL: NCT00723801
Title: Effects of Losartan vs Atenolol on Aortic Stiffness and Diastolic Function in Adults With Marfan Syndrome
Brief Title: Effects of Losartan Versus Atenolol on Aortic and Cardiac Muscle Stiffness in Adults With Marfan Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007p-001762
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Marfan Syndrome
Keywords: Marfan syndrome; Losartan; Atenolol; Diastolic Function; Aortic Stiffness
MeSH Terms: conditions — Marfan Syndrome | interventions — Atenolol; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects Randomized to Losartan (Active Comparator): Losartan: 100 mg PO QD
  Interventions: Drug: Losartan
- Subjects Randomized to Atenolol (Active Comparator): Atenolol: 50 mg PO QD
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Atenolol — Atenolol 50mg PO QD
  Other Names: Tenormin
  Arms: Subjects Randomized to Atenolol
Drug: Losartan — Losartan 100mg PO QD
  Other Names: Cozaar
  Arms: Subjects Randomized to Losartan

SUMMARY:
Marfan syndrome is an inherited connective tissue disorder with morbidity and mortality from aortic dilation and dissection. The degree of aortic dilation and response to beta-blockade (standard of care) vary in adults with Marfan syndrome. However, aortic stiffness is often present, and can be a predictor of aortic dilation and cardiovascular complications. In addition, adults with Marfan syndrome develop left ventricular diastolic dysfunction, which can progress to heart failure. Aortic stiffness and diastolic dysfunction are important and logical therapeutic targets in adults with Marfan syndrome.

TGF-beta mediates disease pathogenesis in Marfan syndrome and contributes to aortic stiffness. The angiotensin receptor blocker, losartan, inhibits TGF-beta activity and reverses aortic wall pathology in a Marfan mouse model. Losartan also decreases aortic stiffness and improves diastolic function in hypertension, renal disease and hypertrophic cardiomyopathy.

This trial is a randomized, double-blind trial of 50 adults with Marfan syndrome, treated with 6 months of atenolol vs. losartan. Arterial tonometry for aortic stiffness and echocardiography for diastolic function will be performed at the beginning and end of treatment. A blood draw for serum markers of extracellular matrix turnover and inflammation will also be performed at 0 and 6 months. We plan to determine whether losartan decreases aortic stiffness and left ventricular diastolic dysfunction significantly more than atenolol.

DETAILED DESCRIPTION:
Please See Summary.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 25 years
* Clinical Marfan Syndrome

Exclusion Criteria:

* Previous aortic or cardiac surgery
* Pregnancy
* Renal Insufficiency
* Medication intolerance

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women;s Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Randomized to Atenolol | Subjects Randomized to Losartan
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Randomized to Atenolol | Subjects Randomized to Losartan | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [25 to 45] | 36 [31 to 44] | 35 [27 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 9 | 16
Pulse wave velocity [Mean (Standard Deviation); unit: meters/second] — Pulse Wave Velocity is a measure of arterial stiffness that is a well-characterized indicator of cardiovascular risk.
  meters/second | 7.5 (1.6) | 7.6 (2.4) | 7.55 (2.0)
Ejection Fraction [Mean (Standard Deviation); unit: %] — Ejection Fraction is a measurement of how much blood volume is ejected from the left ventricle with each contraction. It is a measure of how effectively the heart is pumping blood.
  % | 60 (4) | 62 (6) | 61 (5)

OUTCOME MEASURES:

1. Primary Outcome: Aortic Biophysical Properties - Pulse Wave Velocity
Description: Aortic stiffness was assessed using applanation tonometry (SphygmoCor®, AtCor Medical, West Ryde, NSW, Sydney, Australia) to measure carotid to femoral artery pulse wave velocity (PWV). With the patient lying supine in a quiet environment, a handheld micromanometer-tipped probe was applied to the skin surface over the carotid and femoral arteries, compressing the vessel wall so that transmural forces within the vessel wall were perpendicular to the arterial surface. The distance from the sternal notch to the sites of carotid and femoral pulse acquisition were measured and inputted into the device to represent the relative distance from the carotid to femoral artery. The calculation of distance divided by time of pulse upstroke relative to the upstroke of the QRS on a 3 lead surface EKG was used by the device to calculate velocity. All recorded measurements met the manufacturer's quality control standards integrated into the software package.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: change in meters/second
Arm/Group | Subjects Randomized to Atenolol | Subjects Randomized to Losartan
Number analyzed (Participants) | 17 | 17
change in meters/second | -1.15 (1.68) | -0.22 (.59)

2. Secondary Outcome: Diastolic Function - Ejection Fraction
Description: Two-dimensional echocardiography was performed using a 3.0 MHz transducer (General Electric VIVID 7). Left ventricular and left atrial dimensions were determined in parasternal long axis views. Left ventricular ejection fraction was calculated using the modified Simpsons calculation in the apical two and four chamber views.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Change in % ejection fraction
Arm/Group | Subjects Randomized to Atenolol | Subjects Randomized to Losartan
Number analyzed (Participants) | 17 | 17
Change in % ejection fraction | 1.31 (4.07) | 1.57 (8.29)

ADVERSE EVENTS:
Arm/Group | Subjects Randomized to Atenolol | Subjects Randomized to Losartan
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No